CLINICAL TRIAL: NCT03400410
Title: Hormonal Contraceptive Health Education for Adolescent Males in the Pediatric Emergency Department
Brief Title: Hormonal Contraceptive Health Education for Adolescent Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201706139
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Contraception Behavior
Keywords: Contraception; Education; Male adolescents; Emergency Department; Unintended pregnancy
MeSH Terms: conditions — Contraception Behavior; Emergencies

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator assigned to follow up will be masked to which group a participant was assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Arm (Experimental): This group will take a survey and be asked some sexual history questions including their contraceptive practices with their sexual partner(s). They will then watch the educational video on hormonal contraception and then be asked a few questions about the video. Then they will be asked for an email and phone number for follow up.
  They will then be followed up 3 months from their visit through their contact option of choice (email, text, or call) to take an additional survey with similar sexual history questions and current contraceptive practices including if they have discussed hormonal contraception with their female partners, if their female partners are now using hormonal contraception, and impregnation rates of female partners.
  Interventions: Behavioral: Education Arm
- No Education Arm (No Intervention): This group will take a survey and be asked some sexual history questions including contraceptive practices with their sexual partner(s). They will then be asked for an email and phone number for follow up.
  They will then be followed up 3 months from their visit through their contact option of choice (email, text, or call) to take an additional survey with similar sexual history questions and current contraceptive practices including if they have discussed hormonal contraception with their female partners, if their female partners are now using hormonal contraception, and impregnation rates of female partners.

INTERVENTIONS:
Behavioral: Education Arm — The educational video will be an overview with brief pros and cons of all types of available hormonal contraception. There will be emphasis on the importance of condom use as part of dual method protection.
  Arms: Education Arm

SUMMARY:
Prospective randomized control trial of an educational electronic application on female hormonal contraception for adolescent males in the pediatric emergency department.

DETAILED DESCRIPTION:
Unintended pregnancy among adolescents is a significant public health issue and U.S. adolescents have one of the highest unintended pregnancy rates among industrialized nations. An estimated 9% of male adolescents becoming fathers by the time they are 20 years old. Over 14 million adolescents use emergency departments every year and many of the adolescent males that present to the ED are engaged in high risk sexual behaviors which puts them at high risk for unintended pregnancy. This presents an opportunity to educate males that are at high risk about pregnancy prevention.

This study is a prospective randomized control trial of education about female hormonal contraception for these higher risk adolescent males, 15-21 years old, that present to the Saint Louis Children's Hospital pediatric emergency department. An electronic application will be used to take a sexual history and ask questions about patients' current attitudes and use of hormonal contraception with their partners. They will then be randomized to watch a video on female hormonal contraception (experimental group) or no video (control group). The video will be an overview with brief pros and cons of all available types of hormonal contraception. The app emphasizes importance of condom use as part of dual method protection throughout. All patients will be followed up in 3 months to complete a survey with similar questions on sexual history, discussions with partners, and current contraceptive practices. The hypothesis of the study is that this will lead to increased rates of discussion about hormonal contraception between male adolescents and their sexual partners. This may lead to increased contraceptive use rates and a decrease in unintended pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Male adolescents 15-21 years of age that are sexually active and have ever had vaginal sex that present to the St Louis Children's Hospital pediatric emergency department.

Exclusion Criteria:

* Males that have never had vaginal sex
* Require activation of the trauma system
* Triage as high severity (level 1 or level 2)
* Present for evaluation of abuse, sexual assault, or psychiatric issues
* Unable to speak English
* Wards of the state
* Disabilities that prevent independent use of a tablet device
* Have not completed the electronic adolescent health questionnaire that is standard of care in our emergency department as this is needed for screening purposes

Ages: 15 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — All those that are biologically male, no matter gender identity, that have ever had vaginal sex.
Enrollment: 107 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Discussion rates | 3 months
  Discussion rates of male adolescents with partner(s) about hormonal contraception.

SECONDARY OUTCOMES:
Partner use of hormonal contraception | 3 months
  Partner use of hormonal contraception as assessed by male adolescent.
Fatherhood | Baseline (at initial contact) and 3 months
  Rate of fatherhood of male adolescents in the study.
Male value of partner discussion and hormonal contraceptive knowledge | 3 months
  Yes or No question. Do they believe that partner discussion is important and do they believe that male knowledge of hormonal contraception is important.

CONTACTS AND LOCATIONS:
Overall Officials: Fahd Ahmad, MD, Principal Investigator — Washington Univeristy at St Louis
Locations (1):
- Washington Univeristy at St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] United Nations Population Fund. Adolescent Pregnancy: A Review of the Evidence. 2013; http://www.unfpa.org/publications/adolescent-pregnancy. Accessed Dec 2016, 2016.
- [Background] Centers for Disease Control and Prevention. Reproductive Health: Teen Pregnancy. http://www.cdc.gov/teepregnancy/about/index.htm. Accessed Sept 2016.
- [Background] Mosher WD, Jones J, Abma JC. Intended and unintended births in the United States: 1982-2010. Natl Health Stat Report. 2012 Jul 24;(55):1-28. PMID 23115878
- [Background] Ziv A, Boulet JR, Slap GB. Emergency department utilization by adolescents in the United States. Pediatrics. 1998 Jun;101(6):987-94. doi: 10.1542/peds.101.6.987. PMID 9606224
- [Background] Ahmad FA, Jeffe DB, Plax K, Schechtman KB, Doerhoff DE, Garbutt JM, Jaffe DM. Characteristics of youth agreeing to electronic sexually transmitted infection risk assessment in the emergency department. Emerg Med J. 2018 Jan;35(1):46-51. doi: 10.1136/emermed-2016-206199. Epub 2017 Aug 11. PMID 28801483